CLINICAL TRIAL: NCT01823926
Title: Quantifying Delivery Of Radio Labeled Aerosol During Noninvasive Ventilation To Stable Moderate And Severe Asthmatics: A Randomized, Cross-Over Clinical Trial
Brief Title: Asthma and Quantifying Delivery Of Radio Labeled Aerosol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Daniella Cunha Brandao, PhD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: valdecirtese2
Record Dates: First submitted 2013-03-27; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2012-12

CONDITIONS: Asthma
Keywords: vibrating mesh nebulizers; noninvasive ventilation; residual volume; pulmonary scintigraphy; radioaerosol; nebulization.
MeSH Terms: conditions — Asthma | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): Noninvasive ventilation + jet nebulizer
  Interventions: Other: Noninvasive ventilation; Device: Jet nebulizer
- Experimental Group (Experimental): Noninvasive ventilation + vibrating mesh nebulizer
  Interventions: Other: Noninvasive ventilation; Device: The vibrating mesh nebulizer (VMN)

INTERVENTIONS:
Other: Noninvasive ventilation — Bilevel positive pressure (BiPAP Synchrony, Respironics®, Murrysville, Pennsylvania, USA) was applied through face mask (Comfort Full 2, Respironics®, Murrysville, Pennsylvania, USA) attached with straps and pressure adjusted were 12 cmH2O of inspiratory pressure and 5 cmH2O of expiratory pressure at the beginning of the procedure (França et al., 2006).
Device: Jet nebulizer — Both nebulizers were charged with 2.5 mg of salbutamol and 0.25 mg of ipratropium bromide and 3 mL of saline solution was added to complete 3 Ml. JN (Mist yMax, Air Life, Yorba Linda, USA) was positioned in the circuit using a "T" piece, particle size generation in a 5 µm range (according to the manufacturer information) and flow oxygen tritated at 8 L/min.
  Arms: Control Group
Device: The vibrating mesh nebulizer (VMN) — Both nebulizers were charged with 2.5 mg of salbutamol and 0.25 mg of ipratropium bromide and 3 mL of saline solution was added to complete 3 Ml. VMN (Aeroneb Solo, Galway, Ireland) was positioned in the mask using an elbow (Elbow Kit, Respironics®, Murrysville, Pennsylvania, USA), particle size generation in a 1 µm and connected to electrical energy.
  Arms: Experimental Group

SUMMARY:
Introduction: Inhalation therapy has been established as an efficient route to treat asthma exacerbations, but coupled to noninvasive ventilation (NIV) remains quite challenging.

Objectives: The aim of this study were to compare radiaoaerosol pulmonary index and radioaerosol mass balance in the different compartments (pulmonary and extrapulmonary) using vibrating mesh nebulizers (VMN) and jet nebulizer (JN) coupled to noninvasive ventilation (NIV).

Material and methods: The investigators assessed 10 stable moderate to severe asthmatics in a crossover study. Patients was randomly assigned to participate in both phases of the study: Phase 1(NIV+MN) and phase 2(NIV+JN). DTPA-Tc99m with radioactivity of 25 miC was used to inhaler using JN positioned in the circuit using a "T" piece, particle size generation in a five micron range and oxygen flow tritated at eight L/min and MN was positioned in the mask, particle size generation in a one range and connected to electrical energy. NIV was used a bilevel pressure through a face mask attached with straps and pressure adjusted were 12 cmH2O and 5 cmH2O as inspiratory and expiratory pressures, respectively. After, radioactivity counts were performed using a gama camera and regions of interest were delimited. To calculate aerosol mass balance the investigators considered the amount of radioaerosol deposited into the lungs, upper airways, stomach, nebulizer, circuit, inspiratory and expiratory filters, and mask divided for each of these compartments and represented as a percentage.

ELIGIBILITY:
Inclusion Criteria:

* stable moderate to severe asthma (FEV1 > 60% and > 80% and PEF with a variation of 30% from the predicted values to moderate and FVE1 > 60% and );
* More than one year elapsed since the diagnosis of asthma;
* None exacerbation in the last six months;
* Age between 18 - 60 years, from both sexes,
* Able to understand verbal commands
* Consent to participate in this protocol.

Exclusion Criteria:

* presence of dyspnea;
* smoking history;
* cardiopulmonary diseases (chronic obstructive pulmonary disease, pneumonia, cardiac failure, myocardial infarction, pneumothorax);
* hyperthermia;
* hemodynamic instability (heart rate > 150 bpm and systolic blood pressure < 90 mmHg);
* arrhythmia absence;
* pregnancy
* contraindications for use of noninvasive ventilation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To compare inhaled dose of radioaerosol into the lungs and determine distribution across horizontal and vertical gradients | 10 mouths
  Immediately after inhalation, participants sat in a chair with the back positioned in front to the gamma camera (STARCAM 3200 GE, California, USA) to obtain radioactives counts from the posterior thorax during a period of 500 seconds on a matrix of 256 X 256 matrix. After, participants were positioned sitting in front to the gama camera to obtain images from face. Then, the same procedure was performed to analysis deposition in the nebulizer, circuits, inspiratory filter, expiratory filter and face mask. Counts representing stomach were obtained from posterior thorax and corrections for decay of technetium were used to during extrapulmonary measurements.

SECONDARY OUTCOMES:
To quantify mass balance of the delivery system and different compartments, including intrapulmonary and extrapulmonary deposition. | 10 mouths
  The analysis of deposition in pulmonary and extrapulmonary compartments was expressed as a percentage from the count in each compartment to the total radioaerosol mass generated by nebulizers. The inhaled radioaerosol was considered the sum of deposition into the upper airways, lungs and stomach.

CONTACTS AND LOCATIONS:
Overall Officials: Valdecir G Filho, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Hospital das Clínicas de Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Brandao DC, Lima VM, Filho VG, Silva TS, Campos TF, Dean E, de Andrade AD. Reversal of bronchial obstruction with bi-level positive airway pressure and nebulization in patients with acute asthma. J Asthma. 2009 May;46(4):356-61. doi: 10.1080/02770900902718829. PMID 19484669
- [Result] Galindo-Filho VC, Brandao DC, Ferreira Rde C, Menezes MJ, Almeida-Filho P, Parreira VF, Silva TN, Rodrigues-Machado Mda G, Dean E, Dornelas de Andrade A. Noninvasive ventilation coupled with nebulization during asthma crises: a randomized controlled trial. Respir Care. 2013 Feb;58(2):241-9. doi: 10.4187/respcare.01371. PMID 22781558
- [Result] Soroksky A, Stav D, Shpirer I. A pilot prospective, randomized, placebo-controlled trial of bilevel positive airway pressure in acute asthmatic attack. Chest. 2003 Apr;123(4):1018-25. doi: 10.1378/chest.123.4.1018. PMID 12684289